CLINICAL TRIAL: NCT06555172
Title: Feasibility Trial of a Mindfulness-based mHealth Intervention to Mitigate the Effects of Chronic Workplace Stress Among Juvenile Justice Officers
Brief Title: Feasibility Testing a Meditation App for Professionals Working With Youth in the Legal System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Ashley D Kendall, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-0363
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Anxiety; Depression; Burnout, Professional; Emotion Regulation
MeSH Terms: conditions — Anxiety Disorders; Depression; Burnout, Professional; Emotional Regulation | interventions — Mindfulness; Health Resources

STUDY DESIGN:
Intervention Model Description: Participants will be individually randomized at a 1:1 ratio to 1 of 2 smartphone app conditions: (1) AIM+, a 30-day mindfulness meditation app, or (2) Resource+, a 30-day informational app that is matched to AIM+ for time and structure but provides information on local resources relevant to youth.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action In Mindfulness (AIM)+ (Experimental): Participants randomized to the intervention arm will receive the AIM+ mindfulness meditation app.
  Interventions: Behavioral: Action In Mindfulness (AIM)+
- Resource+ (Active Comparator): Participants randomized to the active control arm will receive the Resource+ informational resource app.
  Interventions: Behavioral: Resource+

INTERVENTIONS:
Behavioral: Action In Mindfulness (AIM)+ — AIM+ is a smartphone-based app that teaches mindfulness meditation to professionals working with legal-involved youth over a 30-day "path." Each day of the path consists of a brief (approximately 5- to 10-minute) audio-guided meditation practice, with brief videos interspersed to illustrate key concepts and promote engagement. In addition to the 30 daily path files, users have access to a menu of "to go" audio-guided meditation practices that they can use as relevant to their workday (e.g., for professionals to listen to before attending a meeting). AIM+ also includes a menu of audio-guided meditation practices that officers can share with the youth on their caseloads (e.g., for youth to listen to before attending court).
  Arms: Action In Mindfulness (AIM)+
Behavioral: Resource+ — Resource+ is a smartphone-based app that is matched to AIM+ for time and structure, but it includes information on community resources that professionals can provide to the youth with whom they work in place of the meditation content featured in AIM+.
  Arms: Resource+

SUMMARY:
This feasibility clinical trial aims to assess the feasibility of implementing a 1-month app-based meditation program with officers in the juvenile legal system and other professionals working directly with legal-involved youth.

DETAILED DESCRIPTION:
Professionals working with legal-involved youth experience high levels of depression, anxiety, and workplace burnout. Mindfulness meditation targets emotion regulation-which appears to be a common mechanism underlying depression, anxiety, and burnout-and it can be effectively delivered via smartphone app. This project will assess the feasibility of implementing a 1-month app-based meditation program with officers and other professionals working with legal-involved youth in Cook County, which houses one of the nation's largest juvenile legal systems. The findings are intended to inform the development of a future, fully-powered hybrid effectiveness-implementation randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Currently working with youth in the juvenile legal system or related juvenile services and programming
* English speaking
* Able to understand and provide consent
* At least 18 years old
* Have an Android or Apple smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
App adherence | 1 month
  Days of objective app usage

SECONDARY OUTCOMES:
Acceptability | 1 month
  Measured by Acceptability of Intervention Measure (AIM). This scale measures acceptability using 4 items, each item rated on a 5-point scale and averaged to yield total scale scores between 1 and 5; higher scores indicate greater acceptability.
Appropriateness | 1 Month
  Measured with the Intervention Appropriateness Measure (IAM). This scale measures appropriateness using 4 items, each item rated on a 5-point scale and averaged to yield total scale scores between 1 and 5; higher scores indicate greater appropriateness.
Feasibility of App Implementation | 1 month
  Measured with the Feasibility of Intervention Measure (FIM). This scale measures feasibility using 4 items, each item rated on a 5-point scale and averaged to yield total scale scores between 1 and 5; higher scores indicate greater feasibility.
Usability | 1 month
  Measured with the System Usability Scale (SUS). This scale measures the usability of products and designs, specifically effectiveness, efficiency, and user satisfaction using 10 items, each item is rated on a 5-point scale; items calculated to produce a total score between 0 and 100; higher scores generally indicate greater usability.
Satisfaction with intervention | 1 month
  Measured with the Client Satisfaction Questionnaire (CSQ-8). This scale measures satisfaction using 8 items, each item is rated on a 4-point scale; total sum scores range from 8 to 32; higher scores indicate higher satisfaction.
Penetration | 1 and 6 month
  Measured via objective app analytics.
  * App analytics track referrals to our clinical trials made by participants through their study app to (a) other officers and (b) youth in the legal system.
  * App analytics track the use by participants of files from their study app that are intended to be shared with youth (i.e., meditation practices to play with youth in the AIM+ app, or resources to be shared with youth in the Resource+ app).

OTHER OUTCOMES:
Anxiety | baseline, 1 month, 6 months
  Measured with the PROMIS Anxiety scale. This scale measures anxiety symptoms over the past week using a computer adaptive test/item bank administers of to 12 items, each rated on a 5-point scale; integrated adaptive scoring yields a T-score and standard error (SE); higher scores indicating more anxiety symptoms.
Depression | baseline, 1 month, 6 months
  Measured with the PROMIS Depression Scale. This scale measures depression symptoms over the past week using a computer adaptive test/item bank administers of to 12 items, each rated on a 5-point scale; integrated adaptive scoring yields a T-score and standard error (SE); higher scores indicating more depression symptoms.
Workplace burnout | baseline, 1 month, 6 months
  Measured with the Maslach Burnout Inventory General (MBI-G). This measure contains three scales measuring emotional exhaustion, depersonalization, and personal accomplishment.
  * The 9-item Emotional Exhaustion (EE) scale assesses feelings of being emotionally overextended and exhausted by one's work, with items rated on a 7-point scale; sum scores range from 0-54; higher scores indicate greater degrees of experienced burnout.
  * The 5-item Depersonalization (DP) scale measures an unfeeling and impersonal response toward recipients of one's service, care, treatment, or instruction, with items rated on a 7-point scale; sum scores range from 0-30; Higher scores correspond to greater degrees of experienced burnout.
  * The 8-item Personal Accomplishment (PA) scale assesses feelings of competence and successful achievement in one's work with people, with items rated on a 7-point scale; sum scores range from 0-48; lower scores correspond to greater degrees of experienced burnout.
Perceived stress | baseline, 1 month, 6 months
  Measured with the Perceived Stress Scale. This scale measures perception of stress over the past month, i.e. the degree to which situations in one's life are appraised as stressful, using 10-items each rated on a 5-point scale; total sum scores range from 0-40, with higher scores indicate more perceived stress.
Anger | baseline, 1 month, 6 months
  Measured with the PROMIS Short Form v1.1 Anger 5a scale. This scale measures anger over the past 7 days using 5 items, each item rated on a 5-point scale; integrated scoring yields a T-score and standard error (SE), with higher scores indicating more anger.
Sleep disturbance | baseline, 1 month, 6 months
  Measured with the PROMIS Short Form v1.0 Sleep Disturbance. This scale measures sleep disturbance over the past 7 days using 8 items, each item rated on a 5-point scale; integrated scoring yields a T-score and standard error (SE); higher scores indicate more sleep disturbance.
Alcohol use | baseline, 1 month, 6 months
  Measured with the PROMIS Short Form v1.0 Alcohol Use 7a. This scale measures alcohol consumption, cravings, or difficulty controlling drinking over the past 30 days using 7 items, each item rated on a 5-point scale; integrated scoring yields a T-score and standard error (SE); higher scores indicate more alcohol consumption, cravings, or difficulty controlling drinking.
Resilience | baseline, 1 month, 6 months
  Measured with the Brief Resilience Scale. This scale measures resilience, i.e. adaptation, thriving, and resistance to illness using 6 items, each item rated on a 5-point scale; averaged to yield total scale scores between 1 and 5; higher scores indicate more resilience.
Mindfulness | baseline, 1 month, 6 months
  Measured with the Five Facets of Mindfulness Questionnaire (FFMQ-15). This scale measures mindfulness with subscales for observing, describing, acting with awareness, non-judging, and non-reactivity using 15 items, each item rated on a 5-point scale; total sum scores range from 15-75; higher scores indicate higher levels of mindfulness.
Regulation of negative mood states | baseline, 1 month, 6 months
  Measured with the Negative Mood Regulation (NMR) Scale. This scale measures regulation of negative mood states using 14 items, each item rated on a 5-point scale; averaged to yield total scale scores between 1 and 5; higher scores indicate a strong belief that one can alter negative moods.
Attentional control | baseline, 1 month, 6 months
  Measured with the Attention Control Scale (ATTC). This scale measures two major components of attention (attention focusing and attention shifting) and consists of 20 items that are rated on a four-point Likert scale from 1 (almost never) to 4 (always); some items are reverse coded and scale scores are calculated as the sum of respective items; higher scores indicate greater attention control.
Current positive and negative mood states | baseline, 1 month
  Measured with the International Positive Affect Negative Affect Schedule Short Form (I-PANAS-SF). This scale measures positive and negative affect, with subscales for positive and negative affect, using 10 items, each item rated on a 5-point scale; sum scores range from 5 to 25; higher scores indicate greater tendency to experiences positive or negative mood, respectively.
Current attentional control | baseline, 1 month
  Measured using 2 items asking about trouble focusing and distraction in the past 3 hours, rated on a scale of 1 (never) to 6 (almost always); items are reverse-coded and averaged to form a composite representing momentary attentional control; higher scores indicate greater attentional control.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be placed in one or more electronic databases which could be used for other research studies
Supporting Information: Study Protocol
Time Frame: Data sharing will generally coincide with publication of the study's main findings and is intended to take place within 1 year after acceptance of the primary manuscripts.
Access Criteria: To be determined

REFERENCES:
- [Derived] Kendall AD, Pela E, Amonica D, Jaworski E, Floyd B; AIM+ Community Advisory Board. Feasibility Testing a Meditation App for Professionals Working With Youth in the Legal System: Protocol for a Hybrid Type 2 Effectiveness-Implementation Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 24;14:e71867. doi: 10.2196/71867. PMID 40273446